CLINICAL TRIAL: NCT06385210
Title: Assessing the Barriers to Surgical Video Recording: a Qualitative Study
Brief Title: Barriers to Routine Surgical Video Recording
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22SM7855
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Minimally Invasive Surgery; Laparoscopic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Semi structured interviews (Experimental): Semi-structured interviews with topic guides centred around the Non adoption, abandonment, scale-up, spread, and sustainability (NASSS) framework will be led by a member of the research team and conducted with all participants. The aim of the interviews is to explore perceived barriers to the uptake of routine surgical video recording. Transcripts will be subsequently thematically analysed using an inductive approach to determine key themes to the barriers of routine surgical video recording.
  Interventions: Other: Semi structured interviews

INTERVENTIONS:
Other: Semi structured interviews — Participants will be interviewed concerning perceived barriers to routine surgical video recording

SUMMARY:
In order to improve the implementation of routine surgical video recording, the researchers want to understand what the challenges associated with the uptake of this technology are. The aim of this study is to explore the barriers faced by key stakeholders including the surgical care team, information governance, and patients within the field of surgical video reporting. The data from this qualitative study will allow the researchers to understand better the challenges associated with uptake of surgical video recording. This will allow the researchers to develop strategies to overcome these challenges and subsequently improve uptake of surgical video recording which will promote safer and more transparent surgery.

DETAILED DESCRIPTION:
This study will involve the use of interviews to determine the barriers to the implementation of surgical video recording.

Participants will be invited to participate in an online 1 on 1 interview 1 on 1. A total of 10-15 participants will be recruited to interview. Interview guides have been developed from the existing literature on the subject. A member of the research team will be present to conduct all interviews. It is estimated that interviews will last between 45-60mins. All interview audio and video will be recorded, as appropriate.

The aim is to recruit 15 participants of which 2-3 will be patient participants and the remaining will be professional participants.

Concerning recruitment of surgical team members: surgeons; trainees; anaesthetists; nursing staff; and operating department practitioners will be invited to participate. Members of the trust's information governance team will also be recruited as key stakeholders within this field as well as representatives from industry who are known personally to the study team.

Non-patient participants will be identified according to their role and be approached directly in person by a member of the study team at their place of work eg outpatient clinic or operating theatres or invited via email for the purposes of recruitment.

Concerning recruitment of patients, appropriate surgical patients satisfying the study inclusion and exclusion criteria will be identified by the direct care team in an outpatient setting through review of patient records. These patients will be under the direct clinical care of members of the study team and will be patients who are awaiting or have recently undergone surgery. The direct care team will explain the rationale of the study and if the potential participant is willing to be contacted, the direct care team will obtain an email address from the potential participant. The potential participant's email address will then be passed on to the study team for further contact.

All interested participants will be emailed a link to an online participant information sheet and consent form.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for professional participants include:

  * Work within the wider surgical care team or in the governance of surgical video or in surgical industry
  * Available to online facilities
  * Explicitly consented Able to understand and communicate in English

Inclusion criteria for patient participants will be as follows:

* Aged 18
* On a waiting list for surgery or have previously undergone surgery in the past 3 years
* Access to online (Teams) facilities
* Explicitly consented Able to understand and communicate in English

Exclusion Criteria:

* Vulnerable adult
* Did not consent to participate
* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Stakeholder perceived barriers to surgical video recording | 6 months
  Participants will undergo a semi-structured interview with topic guides centred around the Non adoption, abandonment, scale-up, spread, and sustainability (NASSS) framework. Interview audio files will be subsequently transcribed and an inductive thematic analysis will be conducted using a grounded-theory approach in order to elucidate key themes to perceived barriers to the uptake of routine surgical video recording.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery and Cancer, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Datasets generated will be available upon reasonable request to the study lead.
Supporting Information: Study Protocol, ICF
Time Frame: 10 years in line with research department data governance guidelines
Access Criteria: Supporting information and datasets generated will be available upon reasonable request to the study lead.